CLINICAL TRIAL: NCT02670187
Title: Phase I, Open-label, Dose Ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of GLS-5300, Administered IM Followed by Electroporation in Healthy Volunteers
Brief Title: Phase I, Open Label Dose Ranging Safety Study of GLS-5300 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 2274
Record Dates: First submitted 2016-01-27; First posted 2016-02-01 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: MERS CoV; MERS-CoV; Middle East Respiratory Syndrome; MERS; DNA Vaccine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GLS-5300 (Experimental): GLS-5300 at 0.67 mg DNA/dose
  Interventions: Biological: GLS-5300
- GLS-5300 at 2 mg DNA/dose (Experimental): GLS-5300 at 2 mg DNA/dose
  Interventions: Biological: GLS-5300
- GLS-5300 at 6 mg DNA/dose (Experimental): GLS-5300 at 6 mg DNA/dose
  Interventions: Biological: GLS-5300

INTERVENTIONS:
Biological: GLS-5300

SUMMARY:
The Middle East Respiratory Syndrome Coronavirus (MERS CoV), a virus related to Severe Acute respiratory syndrome coronavirus (SARS CoV), was first recognized as a cause of severe pulmonary infection in 2012. Infection with MERS CoV has been diagnosed in more than 1600 individuals with a mortality rate between 35% and 40%. GLS-5300 is a DNA plasmid vaccine that expresses the MERS CoV spike (S) glycoprotein. This study will evaluate the safety of GLS-5300 at one of three dose levels following a three-injection vaccination regimen followed by electroporation. The study will also assess immune responses over a 1 year period with respect to the generation of antibody and cellular responses.

DETAILED DESCRIPTION:
GLS-5300 is a DNA plasmid vaccine that expresses the MERS CoV spike (S) glycoprotein. Following administration of the vaccine, a specialized medical device, CELLECTRA®, will deliver brief electrical pulses in a process known as electroporation (EP), to help move DNA into cells more efficiently.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years; military, civilian, male and female.
2. Able to provide consent to participate and having signed an Informed Consent Form.
3. Able and willing to comply with all study procedures.
4. Women of child-bearing potential agree to remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile from enrollment to 3 months following the last injection, or have a partner who is unable to induce pregnancy.
5. Sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception during the study, and agree to continue the use for at least 3 months following the last injection, or have a partner who is permanently sterile or unable to become pregnant;
6. Normal screening ECG or screening ECG with no clinically significant findings;
7. Screening labs must be within normal limits or have only Grade 0-1 findings;
8. No history of clinically significant immunosuppressive or autoimmune disease.
9. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day).
10. Willing to allow storage and future use of samples for MERS CoV related research

Exclusion Criteria:

1. Administration of an investigational compound either currently or within 30 days of first dose;
2. Previous receipt of an investigational product for the treatment or prevention of MERS CoV except if participant is verified to have received placebo;
3. Previous infection with MERS CoV as assessed by self report and solicited exposure history;
4. Administration of any vaccine within 4 weeks of first dose;
5. A BMI greater than or equal to 35;
6. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose;
7. Administration of any blood product within 3 months of first dose;
8. Pregnancy or breast feeding or have plans to become pregnant during the course of the study;
9. History of positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
10. Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
11. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 (CKD Stage II or greater);
12. Baseline screening lab(s) with Grade 2 or higher abnormality;
13. Chronic liver disease or cirrhosis;
14. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
15. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or corticosteroids at a dose less than 20 mg/day);
16. Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
17. Prior major surgery or any radiation therapy within 4 weeks of group assignment;
18. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
19. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD);
20. Metal implants within 20 cm of the planned site(s) of injection;
21. Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection.
22. Prisoner or participants who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
23. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
24. Tattoos covering the injection site area h
25. Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in safety laboratory measures | Day0 through Week 60
Incidence of solicited adverse events after vaccination | Day0 through Week 60
Incidence of unsolicited adverse events after vaccination | Day0 through Week 60
Incidence of serious adverse events | Day0 through Week 60

SECONDARY OUTCOMES:
Binding antibody response to S protein | Day0 through Week 60 following the first dose
Neutralizing antibody response to S protein | Day0 through Week 60 following the first dose
T cell response | Day 0 through Week 60 following the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Kayvon Modjarrad, MD, PhD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Modjarrad K, Roberts CC, Mills KT, Castellano AR, Paolino K, Muthumani K, Reuschel EL, Robb ML, Racine T, Oh MD, Lamarre C, Zaidi FI, Boyer J, Kudchodkar SB, Jeong M, Darden JM, Park YK, Scott PT, Remigio C, Parikh AP, Wise MC, Patel A, Duperret EK, Kim KY, Choi H, White S, Bagarazzi M, May JM, Kane D, Lee H, Kobinger G, Michael NL, Weiner DB, Thomas SJ, Maslow JN. Safety and immunogenicity of an anti-Middle East respiratory syndrome coronavirus DNA vaccine: a phase 1, open-label, single-arm, dose-escalation trial. Lancet Infect Dis. 2019 Sep;19(9):1013-1022. doi: 10.1016/S1473-3099(19)30266-X. Epub 2019 Jul 24. PMID 31351922